CLINICAL TRIAL: NCT02828423
Title: Treatment of Non-contained Infrabony Defects With Enamel Matrix Derivative Alone or in Combination With HA/β-TCP Graft: a 12-month Randomized Controlled Clinical Trial
Brief Title: Regenerative Combined Therapy With Enamel Matrix Derivative and Biphasic Calcium Phosphate Graft
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Universitat Internacional de Catalunya (Other)
Responsible Party: Principal Investigator, Meritxell Losada Martínez, DDS, MS, Associated Professor, Universitat Internacional de Catalunya
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PER-ECL-2011-04-CM
Record Dates: First submitted 2016-06-30; First posted 2016-07-11 (Estimated); Last update posted 2016-07-11 (Estimated); Status verified 2016-07

CONDITIONS: Intrabony Periodontal Defect
Keywords: periodontal regeneration

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control group (Active Comparator): Regeneration therapy of non-contained intrabony defects with enamel matrix derivate (EMD) alone
  Interventions: Procedure: EMD
- Test group (Experimental): Regeneration therapy of non-contained intrabony defects with enamel matrix derivate (EMD) and Biphasic Calcium phosphate (BC)
  Interventions: Procedure: EMD; Procedure: BC

INTERVENTIONS:
Procedure: EMD — Regenerative surgery with EMD
Procedure: BC — Regenerative surgery with BC
  Arms: Test group

SUMMARY:
Background: The use of Enamel Matrix Derivative (EMD) when dealing with non-contained defects may be limited, as EMD does not maintain a space itself. It has been proposed the use of combined therapy, using a bone graft in combination with EMD to avoid the collapse of the flap into the bony defect during the healing time. Therefore the aim of this study is to evaluate the clinical and radiological healing response of non-contained infrabony defects following treatment with a combination of EMD and Biphasic calcium phosphate (BC) or EMD alone.

Methods: Fifty-two patients with at least 1 infrabony defect > 3mm in depth with a probing pocket depth ≥ 6mm were randomly treated with EMD/BC or EMD alone. Clinical and radiographic parameters were evaluated at baseline, 6 and 12 months after surgery. To standardize the procedure an acrylic stent and a millimetre radiographic grid were used. The primary outcome was the change in clinical attachment level (CAL).

Results: Analysis of the data demonstrated a statistically significant difference from baseline within each group (p<0.05), showing a difference in clinical and radiographic parameters at 6 and 12 months for both EMD/BC and EMD alone. However, there were no statistically significant differences between treatment groups.

Conclusions: It was concluded that the treatment of non-contained infrabony defects with EMD, with or without BC, resulted in statistically significant better results after 12 months when compared to baseline measurements. In contrast, the combined approach did not result in a statistically significant improvement.

DETAILED DESCRIPTION:
This is a prospective randomized double blind clinical controlled trial (RCT). Fifty-two systemically healthy adult patients (19 females and 33 males) ranging in age from 35 to 70 years of age, with moderate to advanced chronic periodontitis with at least 1 infrabony defect being >3mm in depth were included. Patients were recruited and treated at the Department of Periodontology dental clinic from the Universitat Internacional de Catalunya, Barcelona, Spain. The sample size calculation was based on a previous pilot study in 10 patients in which differences in between groups where set at 1mm in CAL gain as the primary outcome, with an alpha error of 0.05 and a beta error of 0.9. Thus, the sample size was established for 52 patients including dropouts. The Ethics Committee at the International University of Catalonia (UIC) approved the study design with the code PER-ECL-2011-04-CM. This RCT is registered and follows the CONSORT guidelines as well as the Helsinki declaration for human research. Prior to the initiation of this study, an informed consent was obtained from each patient after explaining the nature of the investigation.

Treatment procedures:

Initial periodontal therapy consisted in oral hygiene instructions until the patient achieved high standards of oral hygiene (modified O'Leary plaque score < 20%), scaling and root planning under local anesthesia and occlusal adjustment if necessary. Four weeks after the completion of phase I therapy, a re-evaluation was performed to confirm the inclusion of the subjects in this clinical research. Probing pocket depth, attachment level, mobility, bleeding on probing and plaque index were assessed. Teeth with mobility greater than class I (Miller 1950) were splinted to adjacent teeth with a twisted wire and light-cured resin.

Before proceeding with the surgical treatment, cast models were obtained from an alginate impression to fabricate an acrylic resin occlusal to standardize clinical measurement with the periodontal probe (Hui-fredy CP-8). The occlusal stent was fabricated using the technique described by Lekovic.

Photographs and standardized reproducible intraoral digital radiographs were obtained from each operated site. The film holder was modified by placing a registration material (Optosil®) on the bite blocks to index the dentition. A paralleling cone technique (7mA-60kV/20ms) was used. A radiopaque millimeter grid was positioned over the radiograph to assess the radiographic measurements. Both the occlusal stent and the radiographic bite blocks with the millimeter grid provided a well-defined and reproducible measurement at each defect and at each examination time point

Clinical and Radiographic parameters:

- Clinical measurements: Two experienced examiners (AP, JN), who were not involved in the surgical procedure, assessed the clinical examinations. A calibration exercise was performed to obtain intra- and inter-examiner reproducibility. According to Polson et al. a training program was followed until reproducibility of 90% was achieved.

The following clinical measurements were taken at the same day of the surgery (baseline) at 6 and 12 months follow-up: 1) Plaque index (PI); 2) Gingival index (GI); 3) Bleeding on probing (BOP); 4) Probing pocket depth (PPD); 5) Gingival recession (GR); 6) Clinical attachment level (CAL) and 7) Mobility (M). PPD, GR and CAL were recorded at the deepest site per tooth: using the same periodontal probe (Hu-friedy CP-8) and a customized stent with guiding grooves.

- Radiographic measurements: The infrabony component was recorded in millimetres. The following measurements were made: 1) distance from the cemento-enamel junction to the bottom of the defect (CEJ-BD), 2) distance from the CEJ to the most coronal extension of the alveolar bone crest (CEJ-BC). The infrabony component (INFRA) of the defects was defined as (CEJ-BD) - (CEJ-BC), 3) angulation of the defect, assessed by measuring the angle between the intersection of a line across the long axis of the tooth and the delimitation of the wall of the defect (GeoGebra® 5.022.0-3D), and 4) number of the remaining walls of the defect, that were confirmed intrasurgically.

Surgical procedures Randomization was performed prior to surgical therapy by a distribution system by sealed cards. One experienced periodontist (AS) performed all surgical procedures instrumented by 2nd and 3rd year periodontal residents (RG, ML). Two different approaches for the treatment of infrabony defects were compared in a randomized controlled double blind clinical trial. Neither the examiners nor the patients were aware of the type of procedure performed. Both surgical procedures were performed under local anaesthesia and the same surgical access to the bony defect was performed. An envelope full thickness mucoperiosteal flap was raised buccal and lingually following simplified papilla preservation incisions. All granulation tissue was removed from the defects and the roots were thoroughly scaled and planed using hand and ultrasonic instruments. The test group was treated by filling the infrabony defect with EMD/BC and the control group with EMD alone. Previously, root surfaces adjacent to all defects were treated with PrefGel® (24% EDTA gel) for 2 minutes according to manufacture's instructions. The root was subsequently rinsed with saline and the bleeding was controlled with the use of gauzes. Topical application of EMD on the root surface in an apical-coronal direction was performed in both study groups. In the test group, the defect was filled in addition with a mixture of the remaining EMD in the syringe and BC. For both treatments, the mucoperiosteal flap was re-positioned and sutured with a non-absorbable suture (Monofilament 6/0) with a horizontal mattress suture and simple suture technique.

Postoperative Care All subjects were instructed to rinse twice daily for 2 weeks with 0,12% clorhexidine gluconate. Tooth brushing and interproximal toothbrush on the regenerated area were initiated at the 15th day after surgical treatment. An analgesic and anti-inflammatory medication were provided for postoperative pain control for 3 days. Antibiotic was provided as well during 7 days. The sutures were removed after 2 weeks, and the surgical sites were gently cleansed with sterile saline using a cotton swab. The patients were scheduled for recall visits on the 1st and 2nd week after surgical treatment and then at 1, 3, 6, and 12 months postoperatively. Oral hygiene was evaluated and supragingival prophylaxis was carried out at each recall visit. Neither probing nor subgingival instrumentation were performed during the first 6 months after surgery.

ELIGIBILITY:
Inclusion Criteria:

* subjects in treatment for periodontal disease with no systemic diseases or conditions that could influence the therapy outcome
* not taking any medication that would affect periodontal healing
* high standards of oral hygiene (PI <20%)
* compliance with the maintenance program
* presence of at least 1 infrabony defect with a probing depth ≥6mm after reevaluation of the hygienic phase and an infrabony component of ≥3mm as detected on radiographs, with any angulation, and exhibiting a 1 or 2 wall intrabony defect
* presence of at least 2mm of keratinized tissue on the buccal aspect of the selected tooth and
* teeth have to be vital or properly treated endodontically.

Exclusion Criteria:

* subjects with any debilitating systemic disease or medication that could affect the periodontium
* heavy smokers (>10 cigarettes/day)
* teeth with class II or III furcation involvement
* mobility > class 2
* strict or predominantly 3-wall defects

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2011-09; Primary Completion 2016-02 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Clinical Attachment Gain | Baseline to 12 months
  Clinical attachment will be recorded in millimeters with a periodontal probe. Differences between baseline and 12 months will be calculated. Measurements will be performed by a masked and calibrated investigator with the aid of a positioning stent over teeth to obtain reproducible measurement in each time point.

SECONDARY OUTCOMES:
Probing pocket depth reduction | Baseline to 12 months
  Probing pocket depth will be recorded in millimeters with a periodontal probe. Differences between baseline and 12 months will be calculated. Measurements will be performed by a masked and calibrated investigator with the aid of a positioning stent over teeth to obtain reproducible measurement in each time point.
Radiograph bone fill gain | Baseline to 12 months
  Radiograph bone fill will be recorded in millimeters with the aid of a millimeter grid positioned over the film when taking the x-ray. Differences between baseline and 12 months will be calculated. Measurements will be performed by a masked and calibrated investigator.

CONTACTS AND LOCATIONS:
Overall Officials: José Nart, PhD, DDS, MS, Study Director — Universitat Internacional de Catalunya

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Losada M, Gonzalez R, Garcia AP, Santos A, Nart J. Treatment of Non-Contained Infrabony Defects With Enamel Matrix Derivative Alone or in Combination With Biphasic Calcium Phosphate Bone Graft: A 12-Month Randomized Controlled Clinical Trial. J Periodontol. 2017 May;88(5):426-435. doi: 10.1902/jop.2016.160459. Epub 2016 Dec 13. PMID 27958765